CLINICAL TRIAL: NCT00006322
Title: Birth Weight Effect on Blood Pressure in Late Childhood
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 925; R01HL060858 (NIH)
Record Dates: First submitted 2000-10-02; First posted 2000-10-03 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2005-03

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension

SUMMARY:
To investigate the relationship of birth weight and childhood blood pressure.

DETAILED DESCRIPTION:
BACKGROUND:

Cardiovascular diseases are the leading causes of morbidity and mortality in the United States. On the basis of an interplay of genetic and environmental factors, these diseases appear to be rooted in childhood. Recent reports implicate the intrauterine nutritional environment regulating fetal growth as a determinant of adult cardiovascular disease. According to this concept, impaired fetal growth, with consequent lower birth weight, results in alteration in organ structure and subsequent functional impairment in later life. Higher blood pressure (BP) has been suggested as the possible link between compromised intrauterine growth and the long-term risk for cardiovascular disease. Despite the many reports which appear to support the low birth weight - high BP hypothesis, this concept is in conflict with the body of data on the association of BP with body size in childhood, adolescence, and adulthood which consistently demonstrates a direct relationship between body weight and BP.

The results of this prospective study contributed an objective body of data to this important issue. If birth measures reflecting intrauterine exposure do contribute significantly to BP in later childhood, then studies focused on the mechanisms regulating this risk are justified. Alternatively, if post-natal/childhood parameters are the major determinants of later BP, then efforts should focus on effective preventive strategies in childhood, such as obesity.

DESIGN NARRATIVE:

To examine the low birth weight - high blood pressure concept, the investigators conducted a prospective study on a cohort of children who were well characterized at birth. In 1988, data on weight, length, BP, gestation and maternal health were obtained on 1,160 newborn cases representing a range of birth weight and gestational age. They re-examined these children at age 11-13 years to test the overall hypothesis that birth weight, as well as other newborn measures of intrauterine growth, did not correlate with BP at age 11-13 years. The aims of the project were to: 1) determine if birth weight contributed to BP and/or body size in childhood; 2) determine if the duration of intrauterine growth in terms of gestational age contributed to BP and body size; 3) determine if newborn ponderal index, a measure of relative fetal growth, contributed to BP and body size; and 4) determine the relative contribution of newborn measures of birth weight, gestational age, BP, ponderal index, and maternal health to BP and body size in late childhood.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Ages: 11 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 1999-07; Study Completion 2003-06 (Actual)

REFERENCES:
- [Background] Falkner B, Hulman S, Kushner H. Effect of birth weight on blood pressure and body size in early adolescence. Hypertension. 2004 Feb;43(2):203-7. doi: 10.1161/01.HYP.0000109322.72948.24. Epub 2003 Dec 15. PMID 14676220